CLINICAL TRIAL: NCT04236271
Title: TELEsurveillance of Patients in PostopErative Bridge surgeryAge CoronairE, Pilot Study
Brief Title: TELEsurveillance of Patients in PostopErative Bridge surgeryAge CoronairE
Acronym: TELE-PEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GFI (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP180485
Record Dates: First submitted 2020-01-10; First posted 2020-01-22 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Bypass
Keywords: connected objects

STUDY DESIGN:
Intervention Model Description: An open, monocentric prospective pilot study evaluating the reliability of post-operative coronary bypass surgery telemonitoring tools and their diagnostic performance for the detection of postoperative complications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient (Experimental): interventional group
  Interventions: Device: connected objects

INTERVENTIONS:
Device: connected objects — a combination of connected devices for measuring physiological parameters and for clinical self-assessment by the patient, for early postoperative coronary bypass surgeries.

SUMMARY:
More than 20,000 patients benefit from coronary bypass surgery in France each year. Median discharge without complication is eight days postoperatively, whereas by day four after surgery, hospitalization is only necessary for medical supervision of the occurrence of complications (scar infection, atrial fibrillation, pericardial effusion), waiting for a downstream bed in cardiac rehabilitation.

Some studies have shown the feasibility of a return home from day 4 after CABG in the United States and England under some conditions of selection and monitoring of patients.

However, there is currently no validated telemonitoring tool for patients in early postoperative coronary bypass surgery.

In this pilot study, during hospitalization for early postoperative coronary bypass surgery, a combination of connected devices for the measurement of physiological parameters and for clinical self-evaluation by the patient will be evaluated. The results of this project will be used as a basis for a future larger study in which an early home discharge can be proposed to patients.

DETAILED DESCRIPTION:
More than 20,000 patients benefit from coronary bypass surgery in France every year. In the case of simple follow-up, the median discharge is eight days postoperatively, whereas by day 4 after surgery, hospitalization is only necessary for medical supervision of the occurrence of complications (scar infection, atrial fibrillation, pericardial effusion), waiting for a downstream bed in cardiac rehabilitation.

Some studies have shown the feasibility of a return home from day 4 after CABG in the United States and England under some conditions of selection and monitoring of patients.

However, there is currently no validated telemonitoring tool for patients in early postoperative coronary bypass surgery.

This is a prospective pilot study, monocentric, open. The intervention consists of the use of connected devices for the monitoring of physiological parameters and functional signs.The use of the connected objects by the patient will take place during hospitalization, in parallel of a standard medical and paramedical follow-up (usual care), from day 4 after coronary bypass a to discharge (or until day 12 maximum, ie 8 days of follow-up).

A combination of connected objects for the measurement of physiological parameters and for clinical self-evaluation by the patient, during early postoperative coronary bypass surgery will be evaluated.

The results of this project will be used as a basis for a future larger study in which an early home discharge can be proposed to patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older at baseline
2. Patient for whom isolated coronary bypass was performed
3. From the 4th day after the operation, epicardial electrodes removed since at least the day before inclusion day, normal blood pressure and heart rate, O2 saturation greater than 94% in ambient air, apyrexia, clean scar, not sign of congestive heart failure
4. From the 4th day after surgery, ECG of the day in sinus rhythm
5. From the 4th day after surgery, hemoglobin> 8g / dl, creatinine clearance> 30ml / min, during a blood sample of less than 24 hours
6. From the 4th day after the operation, no significant abnormalities during a chest X-ray less than 24 hours
7. From the 4th day after surgery, FEVG> 30%, dry pericardium or pericardial effusion ≤ 1cm without compression during transthoracic echocardiography less than 24 hours

Exclusion Criteria:

* Patients at high risk of complications:

  * Insulinorequising diabetics,
  * Non-autonomous,
  * With a context unfavorable to the implementation of the intervention: patient speaking little or no French, patient without social coverage, patient unable to manage complex actions on connected tools.
* Refusal to sign the consent. Protected persons (tutorship, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure measured by connected armband | day 12 postoperatively or discharge from hospital
  The Evolution of blood pressure will be measured daily by connected armband, from day 4 postoperatively to discharge from hospital.
Temperature measured by connected thermometer | day 12 postoperatively or discharge from hospital
  The Evolution of Temperature will be measured daily by connected thermometer, from day 4 postoperatively to discharge from hospital.
Heartbeat measured by connected electrocardiogram | day 12 postoperatively or discharge from hospital
  The heartbeat will be measured daily by connected electrocardiogram, from day 4 postoperatively to discharge from hospital.
scar appearance | day 12 postoperatively or discharge from hospital
  The Evolution of scar appearance will be measured daily by photography, from day 4 postoperatively to discharge from hospital.
pain measured | day 12 postoperatively or discharge from hospital
  The Evolution of pain will be measured daily by an electronic analog visual pain scale, from day 4 postoperatively to discharge from hospital.

SECONDARY OUTCOMES:
Connected armband measurements | day 12 postoperatively or discharge from hospital
  Concordance between connected armband blood pressure measurements, and reference measurements performed by the health care team during hospitalization.
Connected thermometer measurements. | day 12 postoperatively or discharge from hospital
  Concordance between Temperature measured by connected thermometer and reference measurements performed by the health care team during hospitalization disorders, the investigators will evaluate (i) the concordance between the automatic interpretation of the connected ECG and the reading of the classical ECG on the one hand, (ii) the concordance between the automatic interpretation of the ECG connected and re-reading of this same route by a cardiologist.
Connected electrocardiogram | day 12 postoperatively or discharge from hospital
  Concordance between connected electrocardiogram heart rate and reference measurements performed by the health care team during hospitalization. Concerning rhythm disorders, the investigators will evaluate (i) the concordance between the automatic interpretation of the connected ECG and the reading of the classical ECG on the one hand, (ii) the concordance between the automatic interpretation of the ECG connected and re-reading of this same route by a cardiologist.
photography of scar | day 12 postoperatively or discharge from hospital
  Concordance between photography of scar appearance (flow, inflammation), and reference measurements performed by the health care team during hospitalization.
analog visual pain scale | day 12 postoperatively or discharge from hospital
  Concordance between connected an electronic analog visual pain scale and reference measurements performed by the health care team during hospitalization.
Technical failures of connected objects. | day 12 postoperatively or discharge from hospital
  Incidence of occurrence of technical failures of connected objects.
alert algorithms for the diagnosis of postoperative complications | day 12 postoperatively or discharge from hospital
  Sensitivity and specificity of alert algorithms for the diagnosis of postoperative complications (pericardial effusion, heart failure, infection, atrial fibrillation).
Time between surgery and when the patient meets inclusion criteria | day 8 postoperatively
  Time between surgery and when the patient meets the clinical, ECG, biological, radiographic and echocardiographic inclusion criteria
self-measurements performed by the patient | day 12 postoperatively or discharge from hospital
  Proportion of self-measurements performed by the patient using the connected objects among all self-measurements requested.
items completed by the patient in the application | day 12 postoperatively or discharge from hospital
  Proportion of items completed by the patient in the application among the total of items to be completed.
Patient satisfaction | 1 month
  Patient satisfaction measure
Caregiver satisfaction | day 12 postoperatively or discharge from hospital
  Caregiver satisfaction measure
post-operative complications after discharge from hospital | 1 month
  Incidence of occurrence of post-operative complications after discharge from hospital (phone contact on D30).

CONTACTS AND LOCATIONS:
Overall Officials: Claire Cimadevilla, Principal Investigator — APHP
Locations (1):
- Cimadevilla, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided